CLINICAL TRIAL: NCT06451978
Title: You, Me and Nature: A Randomised Pilot Study of a Manualised, Caregiver-led Nature-based Intervention to Improve the Wellbeing of People Living With Mild Cognitive Impairment or Dementia and Their Supporters or Caregivers
Brief Title: You, Me and Nature Pilot Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harmony Jiang (Other)
Responsible Party: Sponsor-Investigator, Harmony Jiang, PhD student, University of Greenwich
Organization: University of Greenwich (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: VCS-FEHHS-02-22
Record Dates: First submitted 2024-05-28; First posted 2024-06-11 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Dementia; Mild Cognitive Impairment
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants will receive the intervention first. Caregivers will attend a one-off training session on how to deliver the intervention. Then the participants will follow the sessions in the intervention manual (8 sessions weekly).
  Interventions: Other: Nature-based intervention
- Waitlist-control group (Active Comparator): Participants will receive the intervention after the intervention group has finished the intervention. Caregivers will attend a one-off training session on how to deliver the intervention. Then the participants will follow the sessions in the intervention manual (8 sessions weekly).
  Interventions: Other: Nature-based intervention

INTERVENTIONS:
Other: Nature-based intervention — The nature-based intervention is a manualised, caregiver-led intervention consisting of a physical manual comprising of 8 sessions of 8 different nature-based activities. It is designed for the person living with dementia or mild cognitive impairment and their caregiver to carry out the sessions together, either in their own home or out in a local area of nature.

SUMMARY:
Background: Nature positively affects people living with dementia. However, there are a lack of nature-based interventions for people living with mild cognitive impairment or dementia who reside in the community.

Aim: This study is testing a caregiver-led nature-based intervention, which has been co-developed with people living with dementia, supporters/caregivers and professionals, and the study design and set-up will also be evaluated. The results will help provide evidence for whether or not to carry out a larger study in the future and will also contribute to the evidence of nature-based interventions for people living with mild cognitive impairment or dementia.

Methods: People from the NHS and charities with a diagnosis of mild cognitive impairment or dementia, and their supporters/caregivers (this pair of participants are called a 'dyad') will be approached. The PhD researcher and dyads will meet to discuss the information sheet, answer any questions, then if they'd like to take part, dyads will each complete a consent form and questionnaire asking about demographics, mental health, and service use. A computer will then randomly assign the dyads into the intervention group or waitlist-control group (who will receive the intervention at the end of the study). Supporters/caregivers in the intervention group will attend a one-off online training session on how to use the manual.

The intervention involves 8 weekly sessions of nature-based activities, including a session evaluation sheet to complete for each session. The PhD researcher will call the supporters/caregivers twice during the intervention to check in. At the end of the intervention, dyads will complete another questionnaire each, and then those in the waitlist-control group will have the opportunity to take part in the intervention. There is also an optional interview that dyads can take part in to talk about their experience of the intervention and the study set-up.

ELIGIBILITY:
Inclusion Criteria:

People living with dementia or mild cognitive impairment (PLWD/MCI)

* Self-reported diagnosis of mild cognitive impairment or dementia (any subtype)
* 18 years old or over
* Has capacity to consent
* Willing to follow the sessions in the manual
* Has a caregiver (family/friend/supporter) that is also willing to take part in the study
* Currently residing in the community (e.g. own home, supported accommodation)
* Sufficient command of English to complete questionnaires and to take part in the intervention

Supporter/caregiver

* An unpaid or informal caregiver, who is caring for a person living with a self-reported diagnosis of mild cognitive impairment or dementia (any subtype) i.e. has at least weekly contact together.
* 18 years old or over
* Has capacity to consent
* The person that they are supporting/caring for is also willing to take part in the study
* Willing to deliver the sessions in the manual
* Willing and able to attend a one-off online caregiver intervention-delivery training session using video conferencing software.
* Currently residing in the community (e.g. own home, supported accommodation)
* Sufficient command of English to complete questionnaires and to deliver the intervention

Exclusion Criteria:

People living with mild cognitive impairment or dementia

1. Currently residing in a nursing or care home
2. Insufficient command of English to complete questionnaires and to take part in the intervention Supporter/caregiver

1. Currently residing in a nursing or care home 2. Insufficient command of English to complete questionnaires and to deliver the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in wellbeing of the person living with dementia or mild cognitive impairment and their caregiver | Post-intervention - 8 weeks after the baseline
  As measured by the Warwick-Edinburgh Mental Well-being Scale (WEMWBS) - 14-item. Minimum score = 14, maximum score = 70. Higher score means better wellbeing (better outcome).

SECONDARY OUTCOMES:
Change in depression of the person living with dementia or mild cognitive impairment and their caregiver | Post-intervention - 8 weeks after the baseline
  As measured by the Patient Health Questionnaire-9 (PHQ-9). Minimum score = 0, maximum score = 27. Higher score means higher levels of depression (worse outcome).
Change in anxiety of the person living with dementia or mild cognitive impairment and their caregiver | Post-intervention - 8 weeks after the baseline
  As measured by the Generalised Anxiety Disorder-7 (GAD-7) Minimum score = 0, maximum score = 21. Higher score means higher levels of anxiety (worse outcome).
Change in connectedness to nature of the person living with dementia or mild cognitive impairment and their caregiver | Post-intervention - 8 weeks after the baseline
  As measured by the Nature Relatedness Scale - 21-item (NR-21). Minimum score = 21, maximum score = 105. Higher score means higher connectedness to nature (neither better or worse outcome).
Change number of medication used and dosages of the person living with dementia or mild cognitive impairment and their caregiver | Post-intervention - 8 weeks after the baseline
  As measured using a non-validated questionnaire which was created by the researchers - this is called 'Medication Use'. The non-validated questionnaire asks for the name of the medication, dosage and dose frequency. No minimum or maximum score. Higher use of medication could mean worse outcome.
Change in number of services used and types of services used by the person living with dementia or mild cognitive impairment and their caregiver | Post-intervention - 8 weeks after the baseline
  As measured using the Client Service Receipt Inventory (CSRI). No minimum or maximum score. Higher use of services could mean better or worse outcome.
Change in cognition score of the person living with dementia or mild cognitive impairment | Post-intervention - 8 weeks after the baseline
  as measured by the Addenbrooke's Cognitive Examination - ACE-III (UK Version A - 2017).
  Minimum score = 0, maximum score = 100. Higher score means higher levels of cognition (better outcome).
Change in positive effects of caregiving score of the caregiver from baseline to post-intervention | Post-intervention - 8 weeks after the baseline
  As measured by the Gain in Alzheimer care Instrument (GAIN). Minimum score = 0, maximum score = 40. Higher score means higher levels of gains in dementia caregiving (better outcome).
Costs of providing the intervention | Post-intervention - 8 weeks after the baseline
  As measured using a non-validated questionnaire. No minimum or maximum score. Higher costs could mean worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Human Sciences, Faculty of Education, Health and Human Sciences, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No